CLINICAL TRIAL: NCT01333124
Title: A Phase 2 Study of Preoperative Chemoradiotherapy With Gemcitabine for Resectable Pancreatic Carcinoma
Brief Title: Preoperative Chemoradiotherapy With Gemcitabine for Resectable Pancreatic Carcinoma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Recruitment delay
Sponsor: National Cancer Center, Korea (Other Government)
Responsible Party: Principal Investigator, Sang-Jae Park, Principal Investigator, National Cancer Center, Korea
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCCCTS-10-500
Record Dates: First submitted 2011-04-01; First posted 2011-04-11 (Estimated); Last update posted 2020-04-06 (Actual); Status verified 2020-04

CONDITIONS: Resectable Pancreatic Carcinoma
Keywords: Preoperative chemoradiotherapy with Gemcitabine
MeSH Terms: interventions — Chemoradiotherapy; Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Radiation: chemoradiotherapy with Gemcitabine (Experimental): Radiation: chemoradiotherapy with Gemcitabine All patients will receive gemcitabine 400 mg/m2 as an intravenous 30-min infusion on day 1, 8, 15, 22, and 29 with radiotherapy.After 4-6 week from end date of chemoradiotherapy, patients undergo preoperative evaluation including CT, PET, CA19-9, CEA. If the patient is feasible for resection on this evaluation, the surgery is performed in 1 to 2 weeks. After surgery, patients will receive gemcitabine 1000 mg/m2 as an intravenous 30-min infusion on day 1, 8, and 15 for every 28 days. Subjects will be treated for at least 1 cycle and to a maximum of four cycles of adjuvant chemotherapy unless there is documented relapse, unacceptable adverse events or withdrawal of consent.
  Interventions: Radiation: chemoradiotherapy with Gemcitabine; Radiation: Radiation: chemoradiotherapy with Gemcitabine

INTERVENTIONS:
Radiation: chemoradiotherapy with Gemcitabine — All patients will receive gemcitabine 400 mg/m2 as an intravenous 30-min infusion on day 1, 8, 15, 22, and 29 with radiotherapy.After 4-6 week from end date of chemoradiotherapy, patients undergo preoperative evaluation including CT, PET, CA19-9, CEA. If the patient is feasible for resection on this evaluation, the surgery is performed in 1 to 2 weeks. After surgery, patients will receive gemcitabine 1000 mg/m2 as an intravenous 30-min infusion on day 1, 8, and 15 for every 28 days. Subjects will be treated for at least 1 cycle and to a maximum of four cycles of adjuvant chemotherapy unless there is documented relapse, unacceptable adverse events or withdrawal of consent.
Radiation: Radiation: chemoradiotherapy with Gemcitabine — Radiation: chemoradiotherapy with Gemcitabine

SUMMARY:
This phase II study is to evaluate the efficacy of preoperative chemoradiotherapy with gemcitabine (400mg/m2, weekly) for resectable pancreatic cancer.

DETAILED DESCRIPTION:
The primary objective of this study is to evaluate the complete (R0) resection rate for patients with and resectable pancreatic cancer treated with preoperative chemoradiotherapy and curative surgery. An experimental arm that result a complete resection rate of at least 90% would merit further study. With 90% power to reject that null hypothesis that the true complete resection rate is ≤75% with a type I error level of 5%, evaluable 53 patients are required. Considering the 20% unevaluable patients due to the immediate distant metastasis after treatment7, 8, 17 and 10% follow up loss, a total of 64 eligible patients will be enrolled.

ELIGIBILITY:
Inclusion Criteria:

* Patients with resectable pancreatic adenocarcinoma
* Age over 18 years old and younger than 70 year old
* Performance status (ECOG scale): 0-1
* Adequate organ functions

  * Hb ≥9.0 g/dl
  * ANC ≥1,500/mm3
  * PLT ≥100,000/mm3
  * Liver function: Total Bilirubin ≤3.0 mg/dl AST/ALT/ALP ≤3× upper limit of normal
  * Creatinine ≤1.5 ULN
* Patients should sign a written informed consent before study entry.

Exclusion Criteria:

* Tumor type other than adenocarcinoma
* Unresectable for resection on preoperative evaluation
* Other primary malignancy (except in situ carcinoma of the cervix or adequately treated basal cell carcinoma of the skin or prior malignancy treated more than 5 years ago without recurrence)
* Prior systemic therapy (for instance, cytotoxic chemotherapy or active/passive immunotherapy)
* Prior radiotherapy
* Major surgery within 4 weeks prior to study treatment
* Serious illness or medical conditions, as follows;

  * congestive heart failure (NYHA class III or IV)
  * unstable angina or myocardial infarction within the past 6 months,
  * significant arrhythmias requiring medication and conduction abnormality such as over 2nd degree AV block
  * uncontrolled hypertension
  * hepatic cirrhosis( ≥ Child class B)
  * interstitial pneumonia, pulmonary adenomatosis
  * psychiatric disorder that may interfere with and/or protocol compliance
  * unstable diabetes mellitus
  * uncontrolled ascites or pleural effusion
  * active infection
* Received any investigational drug or agent/procedure, i.e. participation in another trial within 4 weeks before beginning treatment with study drug
* Pregnant or lactating woman
* Women of child bearing potential not using a contraceptive method
* Sexually active fertile men not using effective birth control during medication of study drug and up to 6 months after completion of study drug if their partners are women of child-bearing potential
* Any patients judged by the investigator to be unfit to participate in the study

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2011-09-28 (Actual); Primary Completion 2017-12-31 (Actual); Study Completion 2017-12-31 (Actual)

PRIMARY OUTCOMES:
Complete resection rate | Within the first 30 days after surgery
  To evaluate the impact of preoperative chemoradiotherapy with gemcitabine by analyzing complete resection rate (R0).

SECONDARY OUTCOMES:
Clinical outcomes | Up to 3years from a initial follow-up
  To investigate the association between radiologic, histopathologic response, complete resection rate of preoperative chemoradiotherapy with gemcitabine and clinical outcomes, such overall survival and disease-free survival.
The association between biomolecular markers and clinical outcomes | Up to 3years until study closed
  To investigate the association between biomolecular markers and clinical outcomes (including tumor response and complete resection rate, etc.)
The feasibility and compliance | Up to 1 year
  To evaluate the feasibility and compliance (acute and late toxicity, esp. gastrointestinal tract toxicity) of preoperative chemoradiotherapy with gemcitabine for resectable pancreatic cancer.

CONTACTS AND LOCATIONS:
Overall Officials: Sang-Jae Park, M.D., Principal Investigator — National Cancer Center, Korea
Locations (1):
- National Cancer Center, Korea, Goyang-si, Gyeonggi-do, South Korea

IPD SHARING:
Plan to Share IPD: No